CLINICAL TRIAL: NCT06524518
Title: Xuanwu Hospital Capital Medical University
Brief Title: A Multicenter Randomized Controlled Study of Interventional Treatment for Operable Stage Ⅱ-Ⅲ Non-small Cell Lung Cancer With Potential Recurrence as Minimal Residual Disease(MRD) Positive
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XuanwuH-NSCLC-MINT
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-06

CONDITIONS: DFS
MeSH Terms: interventions — Immunization

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MRD-negative follow-up (Sham Comparator)
  Interventions: Drug: Chemotherapy combined with immunization
- MRD-positive follow-up (No Intervention)
- MRD-positive adaptive therapy (Experimental)
  Interventions: Drug: Chemotherapy combined with immunization

INTERVENTIONS:
Drug: Chemotherapy combined with immunization — MRD positive patients receive chemotherapy ± immune for 4 cycles before adaptive therapy
  Arms: MRD-negative follow-up; MRD-positive adaptive therapy

SUMMARY:
A prospective, multicenter clinical study designed to explore the efficacy of adaptive therapy based on MRD status in patients with stage II-III non-small cell lung cancer(NSCLC) after treatment. Primary endpoints include 3-year Disease-Free Survival rate (3y-DFS) and median disease-free survival (mDFS).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old
2. gender: men and women can be balanced as far as possible
3. Patients with clinically confirmed stage II-III NSCLC by histopathology have operable conditions
4. no previous exposure to immune-mediated therapy, including but not limited to other anti-CTLA-4, anti-PD-1, anti-PD-L1 And anti-PD-L2 antibodies
5. ECOG behavior status score 0 ~ 1
6. EGFR or ALK driver gene mutation negative
7. organ function level meets the conditions: 1) Hematological examination indicators: absolute neutrophil count (ANC) ≥1.8×109/L, platelet count ≥ 100×109/L, hemoglobin ≥9 g/dL.

2) Appropriate liver function: total bilirubin ≤ 1.5× upper limit of normal (ULN), aspartate aminotransferase (AST), Alanine aminotransferase (ALT) ≤2.5×ULN 3) Appropriate renal function: serum creatinine ≤1.25×ULN, or creatinine clearance ≥60 mL/min

8. Sign informed consent

Exclusion Criteria:

1. Any other anti-tumor treatment before surgery
2. Patients with previous history of other malignant tumors
3. Have a history of interstitial lung disease, drug-induced interstitial disease or any active interstitial lung disease with clinical evidence
4. CT scan at baseline revealed idiopathic pulmonary fibrosis. 4. Pregnant or lactating women
5. multiple lung cancer patients
6. Patient's organ system status:

1) Prior interstitial lung disease, drug-induced interstitial disease, radiation pneumonia or REN requiring hormone therapy Any clinical evidence of active interstitial lung disease 2) In the investigator's judgment, there is a severe or uncontrollable systemic disease (e.g. unstable or uncompensable) Evidence of respiratory, heart, liver or kidney disease) 3) Any unstable systemic disease (including active infection, grade III hypertension, unstable angina, Congestive heart failure, liver, kidney or metabolic disease) 4) Can not accept oral administration, need intravenous high energy nutrition, prior surgery affecting absorption or live Patients with dynamic peptic ulcer

7. Functional level of patients with various organ lesions:

1. Bone marrow: absolute neutrophil count (ANC) < 1.5×109/L, platelets < 90×109/L or blood V1.1 2024.5.29 Albumin < 9 g/dl
2. Liver: serum bilirubin > 1.5 times the upper limit of normal
3. Serum creatinine > 1.25 times the normal value
4. any other disease, neurological or metabolic disorder, the evidence of physical examination or laboratory test results is reasonable Suspected illness or presence of counterindications of use of related drugs or placing subjects at high levels of treatment-related complications The possibility of risk.

8. No R0 resection [ananatomical lobectomy/total pulmonary resection + systemic lymph node dissection (including at least 3 groups of N1) And 3 groups of N2 lymph nodes), both gross and microscopic incisal margins were negative].

9. Situations considered unsuitable for inclusion by other researchers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
DFS | MRD-positive patients were treated 3 years after intervention
  3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, MD,PhD, Study Chair — Capital Medical University
Locations (1):
- Xuanwu Hospital, Beijing, Eijing, China

IPD SHARING:
Plan to Share IPD: No